CLINICAL TRIAL: NCT03080909
Title: Encapsulated Nutrients' Acute Effects on Appetite
Brief Title: Encapsulated Nutrients' Acute Effects on Appetite; ENcapsulated, lipiD, aminO, pRobiotic, SatiEty
Acronym: ENDORSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arne Astrup (Other)
Collaborators: Biocare Copenhagen A/S (Industry)
Responsible Party: Sponsor-Investigator, Arne Astrup, Professor, MD, PhD, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B332
Record Dates: First submitted 2017-02-23; First posted 2017-03-15 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Appetite; Lack or Loss, Nonorganic Origin
Keywords: Satiety; Nutrient; Appetite; Encapsulation; Lipid; Amino acid; Probiotic bacteria

STUDY DESIGN:
Intervention Model Description: A double-blind, randomized crossover design with five arms including four experimental conditions and placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Encapsulated nutients (Active Comparator): Encapsulated nutrients known to be able to stimulate GLP-1 and PYY release. Encapsulated with coating providing release at pH≈7.0 (in the distal part of the ileum) expected to start approximately 3 hour following ingestion.
  The encapsulated nutrients will be provided 30 minutes prior to the standardized fixed breakfast (providing 2000 kJ) and 60 minutes prior to the standardized fixed mid-morning snack (providing 1500 kJ), i.e. test products will be provided 6 hour and 4 hour before the ad libitum test meal, respectively.
  Interventions: Dietary Supplement: Encapsulated nutrients
- Placebo (Placebo Comparator): Nutrients known to have limited stimulation on GLP-1 and PYY release. Encapsulated with coating providing release at pH≈7.0 (in the distal part of the ileum) expected to start approximately 3 hour following ingestion.
  The placebo products will be provided 30 minutes prior to the standardized fixed breakfast (providing 2000 kJ) and 60 minutes prior to the standardized fixed mid-morning snack (providing 1500 kJ), i.e. placebo products will be provided 6 hour and 4 hour before the ad libitum test meal, respectively.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Encapsulated nutrients — Amino acid + Lipid; Probiotic bacteria; Lipid; Amino acid selected on their ability to stimulate release of GLP-1 and PYY
  Arms: Encapsulated nutients
Dietary Supplement: Placebo — Maltodextrin, which is not expected to stimulate release of GLP-1 and PYY
  Arms: Placebo

SUMMARY:
A double-blind, randomized crossover design with five arms including four experimental conditions and placebo will be applied. After having successfully completed screening procedures, eligible participants will be invited to five separate test days. The test days cannot be within the same week, however there is no upper limit for days in between, as long as the participants remain weight stable and do not change diet or physical activity level. Significant changes in diet, physical activity level (evaluated by the sub-investigator) or weight change ±3 kg over the course of the study (from screening to completion of the last test day) results in exclusion of that subject.

DETAILED DESCRIPTION:
For standardization, 48 hours before the test days, the participants will be asked to consume a regular diet compliant to what they usually eat and no excessive alcohol consumption (not above 5 units and no alcohol at all from 8 pm the night before the test days) or intense physical activity compared to what they normally do is allowed. Additionally, the participants must arrive at the study facilities in the morning after an overnight fast (from 10 pm) using non strenuous means of transportation. Furthermore, over the course of the study (from screening (visit 1) to completion of the last test day (visit 6)), the participants are not allowed to change body weight (±3 kg), diet or physical activity level (as judged by the sub-investigator). The participants will be weighed and asked about compliance with additional standardization in a room away from the other participants before initiating each test day. Possible in-compliance with the standardization will be judged by the sub-investigator whether to result in re-scheduling of the visit or to be recorded as a protocol deviation.

Participants arrive at the study facility at 07:30 in the morning. Compliance with standardization is controlled along with registration of possible adverse events, use of concomitant medications and consumption of fermented milk products. During the test days, participants are settled together in an open office, where they are separated at individual tables. During the meals, participants are settled into individual feeding cubicles, where they cannot see each other and are instructed not to talk to each other.

Visual analogue scales (VAS') will be completed for measurement of fasting subjective appetite levels.

The test products (capsules) will be provided 30 minutes prior to a standardized fixed breakfast (providing 2000 kJ) and 60 minutes prior to a standardized fixed mid-morning snack (providing 1500 kJ). An ad libitum test meal will be provided 6 hour after first provision of capsules (time 0). There will be 2 hour interval between the two servings of capsules and 4 hour interval between the second serving of capsules and the ad libitum test meal.

Immediately before and after each episode of capsules and food consumption and at 30 minutes intervals, VAS' will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have provided written informed consent
* Healthy men
* Age between 18 and 60 years
* BMI between 18.5-32 kg/m2
* Regular breakfast eaters (eating breakfast ≥ 4 times a week)

Exclusion Criteria:

* Participants unable to consume or known to get nausea from consuming 20 medium sized capsules (placebo capsules will be provided at screening for test of ability to consume the relevant amount of capsules)
* Participants not able to comply with the study protocol, including consumption of the specific study foods (pictures of study foods shown at screening)
* Any known food allergies or food intolerance likely to affect the present study
* Significant health problems as judged by the principal investigator
* Taking any medication or supplements known to affect appetite or body weight within the past month and/or during the study as judged by the study professional
* Intake of probiotic supplements (any kind of supplements but not including foods containing probiotic) < 4 weeks before study start
* Intake of probiotic supplements (any kind of supplements but not including foods containing probiotic) during the study
* Use of systemic medical treatment likely to interfere with evaluation of the study parameters as judged by the principal investigator
* Smoking, smoking cessation within the past 3 months or nicotine use (electronic cigarettes, gum etc.). Irregular smokers accepted
* Self-reporting currently dieting or having lost/gained significant amount of weight (±3 kg) in the previous 3 months
* Significant weight changes (±3 kg) over the course of the study (from screening to completion of last test day)
* Significant changes in physical activity patterns in the past 4 weeks or significant changes over the course of the study (from screening to completion of last test day) as judged by the sub-investigator
* Significant changes in diet in the past 4 weeks or significant changes over the course of the study (from screening to completion of last test day) as judged by the sub-investigator
* Participants who work in appetite related areas
* Simultaneous or within the past month participating in other clinical trials that can interfere with the study

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Selfreporting
Enrollment: 33 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2017-06-08 (Actual); Study Completion 2017-06-08 (Actual)

PRIMARY OUTCOMES:
Reduced energy intake | up to day 5
  Assessments of ad libitum test meal when exposed to one or more of the encapsulated nutrients compared to the placebo

SECONDARY OUTCOMES:
Subjective appetite sensations | Six hours during each test day between test day 1, 2, 3, 4 and 5 (acute effect)
  Evaluations of each of the subjective appetite sensations assessed by visual analogue scale (VAS) (satiety, fullness, hunger, prospective food consumption, desire to eat)
Subjective appetite sensations in relation to energy consumed | up to day 5
  Assessing the appetite quotient (AQ)

OTHER OUTCOMES:
Subjective nausea assessments | Six hours during each test day between test day 1, 2, 3, 4 and 5 (acute effect)
  VAS assessments for nausea throughout the study test day
Subjective nausea assessments | up to day 5
  End of day questionnaire assessing feeling of nausea after leaving the study facility

CONTACTS AND LOCATIONS:
Overall Officials: Anders Sjödin, MD, PhD, Principal Investigator — Department of Nutrition, Exercise and Sports
Locations (1):
- Department of Nutrition, Exercise and Sports, Copenhagen, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared